CLINICAL TRIAL: NCT03681197
Title: Metformin Use and Clinical Pregnancy Rate in Women With Unexplained Infertility
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elham Raafat (Other)
Responsible Party: Sponsor-Investigator, Elham Raafat, resident of obstetric and gynecology, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1982
Record Dates: First submitted 2018-08-13; First posted 2018-09-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Infertility
Keywords: metformin,unexplained infertility
MeSH Terms: conditions — Infertility | interventions — Metformin; Clomiphene

STUDY DESIGN:
Who Masked: Participant
Masking Description: Each of the consecutive women numbers will be written on sequentially numbered opaque sealed envelope that contains the assignment code.At the time of procedure,the responsible investigator will open the envelope to reveal the assignment,and she will introduce the planned method. Monitoring and follow up will be done. After enrollment,the cases will be randomly allocated into two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin Group (Active Comparator): Will receive metformin plus clomiphene citrate
  Interventions: Drug: Metformin; Drug: Clomiphene Citrate
- Placebo (Placebo Comparator): Will receive placebo plus clomiphene citrate.
  Interventions: Drug: Placebo; Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Metformin — Metformin 850 mg tablet will be started twice daily immediately at booking time and continued with induction by clomiphene citrate, it will be stopped once pregnancy is confirmed.
  Other Names: glucophage
  Arms: Metformin Group
Drug: Placebo — In placebo group,placebo will be strted twice daily at booking time and continued with induction by clomiphene citrate, it will be stopped once pregnancy is confirmed.
  Arms: Placebo
Drug: Clomiphene Citrate — 50 mg of clomiphene citrate will be given starting day 2 of menstrual cycle for 5 days
  Other Names: Clomid

SUMMARY:
The aim of this study is to asses the effect of metformin on clinical pregnancy rate in women with unexplained infertility (randomized controlled trial).

This study will be conducted in infertility clinic,Ain Shams university maternity hospital,170 women with unexplained infertility will be enrolled in this study.

Statistical analysis of the data will be performed .

DETAILED DESCRIPTION:
Metformin is usually used with induction regimen in patients with PCOS as it improves ovulation rate by direct effect on ovarian tissue,Metformin will be used in combination with clomiphene citrate in women with unexplained infertility with previous failed cycle to asses its efficacy on clinical pregnancy rate.

Study will be conducted in infertility clinic,Ain Shams university maternity hospital.Study population comprises women with unexplained infertility aged 20-35 years with total sample size of 170 who willbe randomized into two groups with 85 women in each group.

Group A:is case group who will receive metformin plus clomiphene citrate. Group B:is control group who will receive clomiphene citrate plus placebo. Metformin will be started at time of booking and will be continued till pregnancy is confirmed in a dose of 850 mg twice daily in form of tablet.

Vaginal ultrasound is done for all in day 2 to exclude presence of ovarian cyst and to identify normal appearance of ovaries,then folliculometry on day 9 followed by serial folliculometry every other day till reaching dominant follicle 18 mm or more where HCG intramuscular injection will be given in a dose of 10000 iu .

serum pregnancy test will be done after 16 days. Transvaginal ulterasound will be done on day 35.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-35 years old.
* BMI 20-<30
* FSH 12 IU/L or less
* Normal transvaginal ulterasound(normal uterus and ovaries with no congenital anomalies).
* Patent fallopian tubes assesd by hysterosalpingogram or laparoscopy.
* Normal semen analysis.
* Infertile women with history of previous failed induction cycle.

Exclusion Criteria:

* Women younger than 20 or elder than 35 years old.
* Women with BMI equal to or more than 30.
* Uncorrected congenital or acquired uterine anomaly.
* Other causes of infertility rather than unexplained infertility.
* Patient with Diabetes Mellitus.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | one cycle for each woman (28 days in average)
  Diagnosis of pregnancy by transvaginal ulterasound

CONTACTS AND LOCATIONS:
Overall Officials: Sarah S Moawad, Lecturer, Study Director — Ain Shams Maternity Hospital; Ahmed M Bahaa Eldin, Professor, Study Director — Ain Shams Maternity Hospital; Hisham M Fathy, Professor, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Elham Raafat Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No